CLINICAL TRIAL: NCT03532763
Title: Anti-Inflammatory Effect of Tocotrienol Supplementation in Subjects With Moderately Elevated Inflammation
Acronym: INTOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28701
Record Dates: First submitted 2018-04-26; First posted 2018-05-22 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Inflammation; Cardiovascular Risk Factor
Keywords: Inflammation; Tocotrienols; Cardiovascular disease
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo-controlled, parallel
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocotrienol-rich fraction (Experimental)
  Interventions: Dietary Supplement: Tocotrienol-rich fraction
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tocotrienol-rich fraction — 1 capsule to be taken twice daily after meals for 6 months. Each capsule contains: 200 mg Tocotrienol-rich fraction
  Other Names: Tocovid Suprabio 200 mg
  Arms: Tocotrienol-rich fraction
Dietary Supplement: Placebo — 1 capsule to be taken twice daily after meals for 6 months. Each capsule contains: Palm olein
  Arms: Placebo

SUMMARY:
The objective of this study is to address the anti-inflammatory effect of tocotrienol supplementation in subjects with moderately elevated inflammation.

It is hypothesized that 6 months supplementation of tocotrienols will reduce inflammatory markers of subjects.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, parallel study comparing the effect of tocotrienols vs. placebo will be conducted in subjects with moderately elevated inflammation. Subjects will be supplemented with Tocovid Suprabio 200 mg twice daily or placebo for 6 months. Fasting blood samples will be collected at baseline, 3 months, 6 months. A post-study fasting blood sample will be collected at 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60
* Elevated plasma hs-CRP level of > 1 mg/L < 10 mg/L

Exclusion Criteria:

* Subjects with very high LDL-cholesterol ≥ 4.9 mmol/L
* Subjects with very high hs-CRP level ≥ 10 mg/L
* Pregnancy or lactation
* Current use of vitamin E or corticosteroids
* Significant hepatic and renal impairment
* Fever, cold or infection during bleeding day

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Inflammation | 0, 3, 6, 9 months
  Change in high-sensitivity c-reactive protein (hs-CRP)

SECONDARY OUTCOMES:
Inflammatory markers | 0, 3, 6, 9 months
  Changes in IL-6, IL-1alpha, IL-1beta, TNF-alpha, E-selectin, ICAM-1, VCAM-1
Thrombotic markers | 0, 3, 6, 9 months
  Changes in PAI-1, D-dimer
Lipid profile | 0, 3, 6, 9 months
  Changes in TC, LDL, HDL, ApoA1, ApoB
Glucose homeostasis | 0, 3, 6, 9 months
  Changes in Glucose, insulin, c-peptide

CONTACTS AND LOCATIONS:
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia